CLINICAL TRIAL: NCT03536806
Title: Clinical Efficacy of Potassium Canrenoate - Canrenone in Sinus Rhythm Restoration Among Patients With Atrial Fibrillation and Elevated Blood Pressure - a Pilot Randomized Controlled Trial.
Brief Title: Clinical Efficacy of Potassium Canrenoate in Sinus Rhythm Restoration Among Patients With Atrial Fibrillation.
Acronym: CANREN-AF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Principal Investigator, Rafał Dąbrowski, Rafal Dabrowski, MD, PhD, National Institute of Cardiology, Warsaw, Poland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2.62/VII/16
Record Dates: First submitted 2018-05-12; First posted 2018-05-25 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Atrial Fibrillation, Paroxysmal
Keywords: Pharmacological cardioversion; Canrenone
MeSH Terms: conditions — Atrial Fibrillation | interventions — Sodium Chloride; Canrenone

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Comparator: Placebo (Placebo Comparator): Any patient fulfilling the inclusion criteria will be prepared to pharmacological cardioversion in a standard way comprising of standard baseline 12-lead ECG, continuous ECG monitoring, periodic noninvasive blood pressure monitoring (BP) and iv line. Patients assigned to control group will be administered saline 0.9% in bolus of 10 cm3 within 2-3 minutes. After drug administration the patient will be observed for 2 hours after the last dose with exit ECG and BP measure taken at the end of observation. Further treatment of the patient will depend on clinical condition and will follow appropriate clinical guidelines.
  Interventions: Drug: Saline 0.9%
- Experimental: canrenone (Experimental): Any patient fulfilling the inclusion criteria will be prepared to pharmacological cardioversion in a standard way comprising of standard baseline 12-lead ECG, continuous ECG monitoring, periodic noninvasive blood pressure monitoring (BP) and iv line. After administration of canrenone: dose 200 mg (1 ampule a 10 ml) within 2-3 minutes the patient will be observed for 2 hours after the dose with exit ECG and BP measure taken at the end of observation.
  Interventions: Drug: Canrenone

INTERVENTIONS:
Drug: Saline 0.9% — Patients assigned to control group will be administered saline 0.9% in bolus of 10 cm3 within 2-3 minutes. BP will be measured before injection.
  Other Names: saline 0.9% in bolus of 10 cm3
  Arms: Placebo Comparator: Placebo
Drug: Canrenone — Patients assigned to canrenone group will be administered canrenone in bolus of 200 mg diluted to 10 cm3 within 2-3 minutes in one dose. Drug administration will be stopped in case of serious adverse event. Further treatment of the patient will depend on clinical condition and will follow appropriate clinical guidelines.
  Other Names: canrenone in bolus of 200 mg diluted to 10 cm3
  Arms: Experimental: canrenone

SUMMARY:
The purpose of this randomized, double blind, placebo-controlled, superiority clinical trial was to assess clinical efficacy of potassium canrenoate - canrenone in rapid conversion of atrial fibrillation to sinus rhythm.

DETAILED DESCRIPTION:
Canrenone is a specific antagonist of aldosterone. It is a competitive inhibitor of aldosterone receptors and inhibits the effects of aldosterone. Spironolactone is a prodrug which is active after its conversion into canrenone. By inhibiting the effects of aldosterone it increases aqueous and sodium diuresis and is classified as a diuretic. It decreases urinary elimination of potassium and increases urinary excretion of calcium. Canrenone is used for the treatment of primary or secondary hyperaldosteronism, edema and ascites of congestive heart failure and cirrhosis, and in the treatment of the arterial hypertension. Current evidence supports renin-angiotensin-alodsterone (RAAS) inhibition: angiotensin-converting-enzyme inhibitors (ACE-I), angiotensin receptor blockers (ARB) or, potentially, mineralocorticoid receptor antagonists (MRA) as an upstream therapy for atrial fibrillation (AF) management. It has been demonstrated that plasma aldosterone concentration may be increased in patients with AF episode, and it lowers after cardioversion. Only canrenone (potassium canrenoate) may be administered intravenously. Canrenone increases plasma level of potassium, lowers blood pressure and reduces preload at the same time.

To show superiority of canrenone over placebo a sample size of 80 patients was calculated based on following assumptions: two-tailed test, a type I error of 0.01, a power of 90%, efficacy of placebo 5%, efficacy of canrenone 50% and 20% drop-out rate to fulfill the criteria of intention-to-treat analysis. Due to presumed lack of statistical power the secondary end points and safety endpoints will be considered exploratory.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent for enrolment
* patients aged between 40 and 75 years
* atrial fibrillation episode lasting for less than 48 hours, documented by the ECG
* potassium plasma levels < 4.5 mmol/l
* blood pressure > 120/80 mmHg
* stable cardiopulmonary status (according to attending physician's assessment)
* in case of left ventricle injury suspicion or unclear medical history of cardiac insufficiency, enrolment will be possible after echocardiographic examination

Exclusion Criteria:

* no written informed consent for enrollment
* allergy to canrenone
* cardiac insufficiency or LVEF (left ventricular ejection fraction) < 40%
* systolic BP < 120/80 mmHg
* history of canrenone treatment in the 30 days before enrollment
* average QRS rate > 160 p.m.
* advanced hepatic or renal failure
* history of acute coronary syndrome, CABG (coronary artery bypass grafting), TIA (transient ischemic attack) or stroke within the previous 30 days
* pre-excitation syndrome (which has not been treated with accessory pathway ablation).
* atrial fibrillation due to a valvular heart disease
* atrial fibrillation episode resulting in myocardial ischemia (chest pain, ischemic changes in the ECG)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Conversion of atrial fibrillation to sinus rhythm. | Time Frame: 2 hours.
  Conversion of atrial fibrillation to sinus rhythm confirmed in standard 12-lead ECG during observation period after first iv bolus.

SECONDARY OUTCOMES:
Time to conversion of atrial fibrillation to sinus rhythm. | Time Frame: 2 hours.
  Time to conversion of atrial fibrillation to sinus rhythm in minutes since injection.
Atrial fibrillation recurrence within observation period. | Time Frame: 2 hours.
  Atrial fibrillation recurrence within observation period.
Serious adverse reactions. | Time Frame: 24 hours.
  Serious adverse reactions, which refer to every event requiring admission to a hospital or extended observation.
Safety outcome (exploratory analysis). | Time Frame: 24 hours.
  hypotension < 90 mm Hg, cardiac conduction abnormalities, new arrhythmia occurrence, other

CONTACTS AND LOCATIONS:
Overall Officials: Rafał Dąbrowski, MD, PhD, Principal Investigator — Institute of Cardiology; Tomasz Hryniewiecki, MD, PhD, Study Chair — Institute of Cardiology

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dabrowski R, Segiet-Swiecicka A, Sawicki S, Kowalik I, Jaworski K, Farkowski M, Kubaszek-Kornatowska A, Michalek P, Dluzniewski M, Szwed H, Hryniewiecki T, Karwowski J; CANREN-AF investigators. Clinical Efficacy of Canrenone in Restoring Sinus Rhythm in Patients With Atrial Fibrillation-A Pilot, Randomized, Double-Blind Study. J Cardiovasc Pharmacol Ther. 2025 Jan-Dec;30:10742484251356361. doi: 10.1177/10742484251356361. Epub 2025 Jul 29. PMID 40734383
- [Derived] Dabrowski R, Syska P, Maczynska J, Farkowski M, Sawicki S, Kubaszek-Kornatowska A, Michalek P, Kowalik I, Szwed H, Hryniewiecki T. Clinical efficacy of potassium canreonate-canrenone in sinus rhythm restoration among patients with atrial fibrillation - a protocol of a pilot, randomized, double -blind, placebo-controlled study (CANREN-AF trial). Trials. 2020 May 12;21(1):397. doi: 10.1186/s13063-020-04277-3. PMID 32398047